CLINICAL TRIAL: NCT03735121
Title: A Randomized, Multicenter, Phase Ib/III Study to Investigate the Pharmacokinetics, Efficacy, and Safety of Atezolizumab Subcutaneous Compared With Atezolizumab Intravenous in Patients With Previously Treated Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study to Investigate Atezolizumab Subcutaneous in Patients With Previously Treated Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP40657; 2018-002328-18 (EudraCT Number)
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Results first posted 2023-06-13 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: Intervention study model can be sequential or in parallel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Atezolizumab (Part 2) (Experimental): Atezolizumab
  Interventions: Drug: Atezolizumab
- Cohort 1: Atezolizumab+rHuPH20 (Part 1) (Experimental): Atezolizumab+recombinant human hyaluronidase (rHuPH20), followed by Atezolizumab
  Interventions: Drug: Atezolizumab; Drug: rHuPH20
- Cohort 2: Atezolizumab+rHuPH20 (Part 1) (Experimental): Atezolizumab+rHuPH20, followed by Atezolizumab
  Interventions: Drug: Atezolizumab; Drug: rHuPH20
- Cohort 3: Atezolizumab+rHuPH20(Part 1) (Experimental): Atezolizumab+rHuPH20, followed by Atezolizumab
  Interventions: Drug: Atezolizumab; Drug: rHuPH20
- Atezolizumab + rHuPH20 (Part 2) (Experimental): Atezolizumab + rHuPH20
  Interventions: Drug: Atezolizumab; Drug: rHuPH20

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered as per the schedule specified in arm or cohort.
  Other Names: Tecentriq
Drug: rHuPH20 — rHuPH20 will be administered as per the scheduled specified in the cohort for Part 1.
  Other Names: ENHANZE
  Arms: Atezolizumab + rHuPH20 (Part 2); Cohort 1: Atezolizumab+rHuPH20 (Part 1); Cohort 2: Atezolizumab+rHuPH20 (Part 1); Cohort 3: Atezolizumab+rHuPH20(Part 1)

SUMMARY:
This study will evaluate the pharmacokinetics, safety, and efficacy of atezolizumab subcutaneous (SC) compared with atezolizumab intravenous (IV) in participants with locally advanced or metastatic Non-Small Cell Lung Cancer (NSCLC) who have not been exposed to cancer immunotherapy (CIT) and for whom prior platinum-based therapy has failed. The study is comprised of two parts, as follows: A dose-finding part (Part 1, Phase Ib) will aim to identify the dose of atezolizumab SC to be tested in Part 2. A dose-confirmation part (Part 2, Phase III, randomized) will aim to confirm that the dose moved forward from Part 1 yields drug exposure that is comparable to that of atezolizumab IV.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented locally advanced or metastatic NSCLC
* Prior platinum-containing regimen or disease recurrence ≤ 6 months since prior platinum-based adjuvant/neoadjuvant regimen.
* Measurable disease as defined by RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy ≥12 weeks
* Adequate hematologic and end-organ function

Additional Inclusion Criteria (Part 2 Only) • Availability of tissue and known epidermal growth factor receptor (EGFR) status

Exclusion Criteria:

* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* Uncontrolled or symptomatic hypercalcemia
* Pregnancy or breastfeeding
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis
* Severe infection ≤ 4 weeks
* Treatment with therapeutic oral or IV antibiotics ≤ 2 weeks prior to study treatment
* Significant cardiovascular disease
* Prior allogeneic stem cell or solid organ transplantation
* Treatment with a live, attenuated vaccine ≤ 4 weeks
* Treatment with systemic immunostimulatory agents ≤ 4 weeks or 5 half-lives of the drug
* Treatment with systemic immunosuppressive medication ≤ 2 weeks

Additional Exclusion Criteria (Part 2 Only)

• Tested tumor programmed death-ligand-1 (PD-L1) expression status with an intention to treat the patient if positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2024-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (74):
- Argentina (3):
  - Fundación CENIT para la Investigación en Neurociencias, Buenos Aires
  - Centro Oncologico Riojano Integral (CORI), La Rioja
  - Consultorio Dr. Miguel Angel Escudero, Salta
- Brazil (4):
  - Oncosite - Centro de Pesquisa Clinica Em Oncologia Ltda, Ijuí, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - INCA 1- Instituto Nacional de Câncer X, Rio de Janeiro
- Chile (3):
  - Bradford Hill Centro de Investigaciones Clinicas, Recoleta
  - James Lind Centro de Investigación Del Cáncer, Temuco
  - Oncocentro Apys, Viña del Mar
- China (5):
  - Jilin Cancer Hospital, Changchun
  - West China Hospital - Sichuan University, Chengdu
  - Sir Run Run Shaw Hospital Zhejiang University, Hangzhou
  - Jinan Central Hospital, Jinan
  - Henan Cancer Hospital, Zhengzhou
- Costa Rica (2):
  - Clinica CIMCA, San José
  - ICIMED Instituto de Investigación en Ciencias Médicas, San José
- France (2):
  - APHM, Marseille
  - Ico Rene Gauducheau, Saint-Herblain
- Greece (2):
  - General Hospital "G.Papanikolaou", Asvestochóri
  - Sotiria Hospital, Athens
- Guatemala (4):
  - INTEGRA Cancer Institute, Guatemala City
  - Oncomedica, Guatemala City
  - Grupo Angeles, Guatemala City
  - Hospital El Pilar, Guatemala City
- Hungary (2):
  - Matrai Gyogyintezet, Mátraháza
  - Református Pulmonológiai Centrum, Törökbálint
- Italy (2):
  - Asst Papa Giovanni XXIII, Bergamo, Lombardy
  - IRCCS Istituto Clinico Humanitas, Rozzano, Lombardy
- Riga East Clinical University Hospital Latvian Oncology Centre, Riga, Latvia
- Mexico (2):
  - Health Pharma Professional Research, Mexico City, Mexico CITY (federal District)
  - Cuidados oncologicos, Querétaro City, Querétaro
- New Zealand (4):
  - Auckland City Hospital, Cancer and Blood Research, Auckland
  - Christchurch Clinical Studies Trust Ltd, Christchurch
  - Waikato Hospital - Cancer and Blood Research Trials Unit, Hamilton
  - Tauranga Hospital, Clinical Trials Unit, Tauranga
- Peru (4):
  - Centro Medico Monte Carmelo, Arequipa
  - Clínica San Gabriel, Lima
  - Oncosalud Sac, Lima
  - Clinica Internacional, Sede San Borja, Lima
- Poland (4):
  - Regionalny Szpital Specjalistyczny im. W. Bieganskiego, Grudzi?dz
  - Centrum Terapii Wspolczesnej, Lodz
  - Mazowieckie Centrum Leczenia Chorob Pluc i Gruzlicy, Otwock
  - Narodowy Instytut Onkologii im. M. Sklodowskiej-Curie, Warsaw
- Russia (8):
  - Chelyabinsk Regional Clinical Oncology Dispensary, Chelyabinsk, Moscow Oblast
  - FSBI Russian Oncology Research Center n.a. Blokhin of MOH RF, Moscow, Moscow Oblast
  - MEDSI Clinical Hospital on Pyatnitsky Highway, Moscow, Moscow Oblast
  - Filial #1 Regional Oncology Dispensary of Nizhniy Novgorod, Nizhny Novgorod, Niznij Novgorod
  - Mordovia State University, Saransk, Respublika Mordoviya
  - SBIH Kaluga Region Clinical Oncology Dispensary, Kaluga
  - Murmansk Regional Clinical Hospital named after P.A. Bayandin, Murmansk
  - Multidisciplinary clinic Reaviz, Samara
- South Africa (3):
  - Groote Schuur Hospital ( Uni of Capetown ), Cape Town
  - Wilgers Oncology Centre, Pretoria
  - Sandton Oncology Medical Group, Sandton
- South Korea (2):
  - Asan Medical Center, Seoul
  - Samsung Medical Centre, Seoul
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
- Thailand (8):
  - Vajira Hospital, Bangkok
  - Chulalongkorn Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Faculty of Med. Siriraj Hosp., Bangkok
  - Prapokklao Hospital, Chanthaburi
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Prince of Songkla University, Hat Yai
  - Udonthani Cancer Hospital, Udonthani, Muang,Udonthani
- Turkey (Türkiye) (2):
  - Medipol University Medical Faculty, Istanbul
  - Ege Uni Medical Faculty Hospital, Izmir
- Ukraine (4):
  - Municipal Institution City Clinical Hospital #4 of Dnipro City Council, Dnipropetrovsk, Katerynoslav Governorate
  - Communal Non profit Enterprise Regional Center of Oncology, Kharkiv, Kharkiv Governorate
  - Ivano-Frankivsk Regional Oncology Center, Ivano-Frankivsk
  - RCI Sumy Regional Clinical Oncological Dispensary, Sumy
- Birmingham Heartlands Hospital, Birmingham, United Kingdom

REFERENCES:
- [Derived] Burotto M, Zvirbule Z, Mochalova A, Runglodvatana Y, Herraez-Baranda L, Liu SN, Chan P, Shearer-Kang E, Liu X, Tosti N, Zanghi JA, Leutgeb B, Felip E. IMscin001 Part 2: a randomised phase III, open-label, multicentre study examining the pharmacokinetics, efficacy, immunogenicity, and safety of atezolizumab subcutaneous versus intravenous administration in previously treated locally advanced or metastatic non-small-cell lung cancer and pharmacokinetics comparison with other approved indications. Ann Oncol. 2023 Aug;34(8):693-702. doi: 10.1016/j.annonc.2023.05.009. Epub 2023 Jun 1. PMID 37268157
- [Derived] Felip E, Burotto M, Zvirbule Z, Herraez-Baranda LA, Chanu P, Kshirsagar S, Maiya V, Chan P, Pozzi E, Marchand M, Monchalin M, Tanaka K, Tosti N, Wang B, Restuccia E. Results of a Dose-Finding Phase 1b Study of Subcutaneous Atezolizumab in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer. Clin Pharmacol Drug Dev. 2021 Oct;10(10):1142-1155. doi: 10.1002/cpdd.936. Epub 2021 Mar 31. PMID 33788415

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 438 participants with previously treated locally advanced or metastatic non-small cell lung cancer (NSCLC) who were cancer immunotherapy (CIT)-naïve and for whom prior platinum-based therapy failed took part in the study across 23 countries from 27 December 2018 to 22 November 2024. The study is considered "Completed" because all the pre-planned study activities and analyses have been performed.
Pre-assignment Details: Study consisted of 2 parts: Part 1 (Dose Finding) & Part 2 (Dose Confirmation). Health care professionals (HCPs) who administered the study treatment to participants were not enrolled in the study. To evaluate the HCPs' reported experience with administration of atezolizumab SC & atezolizumab IV, the HCPs were asked to complete two questionnaires: 'HCP SC Versus IV Perspective' & 'HCP SC Perspective'.
  No data other than the HCP's responses to these Questionnaires were collected in this study.
Groups:
- Part 1 Cohort 1: Atezolizumab SC Co-mix 1800 mg: Participants received atezolizumab, 1800 milligrams (mg), co-mixed with rHuPH20, as SC injection on Cycle 1 Day 1 (1 cycle=21 days), followed by atezolizumab, 1200 mg, as an IV infusion, every 3 weeks (Q3W) on Day 1 of subsequent cycles (1 cycle=21 days) until disease progression (PD), loss of clinical benefit, unacceptable toxicity, or withdrawal of consent.
- Part 1 Cohort 2: Atezolizumab SC Co-mix 1200 mg: Participants received atezolizumab, 1200 mg, co-mixed with rHuPH20, as SC injection, Q2W, on Day 1 of the first 3 cycles (Cycle 1-3=14 days), followed by atezolizumab, 1200 mg, as an IV infusion, Q3W, on Day 1 of subsequent cycles (1 cycle=21 days) until PD, loss of clinical benefit, unacceptable toxicity, or withdrawal of consent.
- Part 1 Cohort 3: Atezolizumab SC Co-mix 1800 mg: Participants received atezolizumab, 1800 mg, co-mixed with rHuPH20, as SC injection, Q3W, on Day 1 of first 3 cycles, followed by atezolizumab, 1200 mg, as an IV infusion, Q3W on Day 1 for subsequent cycles (1 cycle=21 days) until PD, loss of clinical benefit, unacceptable toxicity, or withdrawal of consent.
- Part 2: Atezolizumab IV 1200 mg: Participants received atezolizumab, 1200 mg, as an IV infusion, Q3W, on Day 1 of each cycle (1 cycle=21 days) until PD, loss of clinical benefit, or unacceptable toxicity.
- Part 2: Atezolizumab SC 1875 mg: Participants received atezolizumab, 1875 mg, co-formulated with rHuPH20, as SC injection, on Day 1 of each cycle (1 cycle=21 days) until PD, loss of clinical benefit, or unacceptable toxicity.
Period: Overall Study
Arm/Group | Part 1 Cohort 1: Atezolizumab SC Co-mix 1800 mg | Part 1 Cohort 2: Atezolizumab SC Co-mix 1200 mg | Part 1 Cohort 3: Atezolizumab SC Co-mix 1800 mg | Part 2: Atezolizumab IV 1200 mg | Part 2: Atezolizumab SC 1875 mg
Started | 13 | 15 | 39 | 124 | 247
Completed | 8 | 7 | 13 | 0 | 0
Not Completed | 5 | 8 | 26 | 124 | 247
Not completed — Death | 3 | 6 | 19 | 97 | 205
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 3
Not completed — New Therapy | 0 | 1 | 0 | 0 | 0
Not completed — Study Ended by Sponsor | 1 | 0 | 1 | 17 | 28
Not completed — Withdrawal by Subject | 1 | 1 | 6 | 8 | 11

BASELINE CHARACTERISTICS:
Population: Part 1: Intent-to-treat (ITT) population included all enrolled participants. Part 2: Full analysis set (FAS) included all participants who were randomized with participants grouped per their assigned treatment.
  HCPs who administered the study treatment to participants were not enrolled in the study. To evaluate the HCPs' reported experience with administration of atezolizumab SC & IV, the HCPs were asked to complete 2 questionnaires. No baseline data were collected for the HCPs in this study.
Groups:
- Part 1 Cohort 1: Atezolizumab SC Co-mix 1800 mg: Participants received atezolizumab, 1800 mg, co-mixed with rHuPH20, as SC injection on Cycle 1 Day 1 (1 cycle=21 days), followed by atezolizumab, 1200 mg, as an IV infusion, Q3W on Day 1 of subsequent cycles (1 cycle=21 days) until PD, loss of clinical benefit, unacceptable toxicity, or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohort 1: Atezolizumab SC Co-mix 1800 mg | Part 1 Cohort 2: Atezolizumab SC Co-mix 1200 mg | Part 1 Cohort 3: Atezolizumab SC Co-mix 1800 mg | Part 2: Atezolizumab IV 1200 mg | Part 2: Atezolizumab SC 1875 mg | Total
Number analyzed (Participants) | 13 | 15 | 39 | 124 | 247 | 438
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 19 | 58 | 137 | 229
  >=65 years | 5 | 8 | 20 | 66 | 110 | 209
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 12 | 42 | 72 | 140
  Male | 5 | 9 | 27 | 82 | 175 | 298
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 9 | 15 | 24
  Asian | 2 | 2 | 1 | 33 | 47 | 85
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 2 | 1 | 3
  Black or African American | 0 | 0 | 0 | 1 | 2 | 3
  White | 8 | 11 | 36 | 74 | 174 | 303
  More than one race | 0 | 0 | 0 | 5 | 6 | 11
  Unknown or Not Reported | 3 | 2 | 2 | 0 | 2 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 12 | 36 | 61 | 115
  Not Hispanic or Latino | 9 | 7 | 25 | 88 | 185 | 314
  Not Stated | 3 | 3 | 2 | 0 | 0 | 8
  Unknown | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Serum Trough Concentration (Ctrough) of Atezolizumab at Cycle 1
Time Frame: Pre-dose on Day 1 of Cycle 2 (Cycle length=21 days for cohorts 1 and 3 and 14 days for cohort 2)
Population: Pharmacokinetic (PK)-evaluable population included all participants who received at least one dose of atezolizumab and had at least 1 evaluable post dose PK sample that could affect PK results. Overall number analyzed is the number of participants with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Part 1 Cohort 1: Atezolizumab SC Co-mix 1800 mg | Part 1 Cohort 2: Atezolizumab SC Co-mix 1200 mg | Part 1 Cohort 3: Atezolizumab SC Co-mix 1800 mg
Number analyzed (Participants) | 13 | 15 | 35
micrograms per milliliter (μg/mL) | 121 (42.8) | 77.5 (51.4) | 78.3 (88.6)

2. Primary Outcome: Part 2: Observed Serum Ctrough of Atezolizumab at Cycle 1
Time Frame: Predose on Day 1 of Cycle 2 (Cycle length =21 days)
Population: Per Protocol PK evaluable population included all participants randomized to the atezolizumab SC and atezolizumab IV treatment arms who did not have protocol deviations that could affect Cycle 1 observed Ctrough results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 2: Atezolizumab IV 1200 mg | Part 2: Atezolizumab SC 1875 mg
Number analyzed (Participants) | 97 | 205
μg/mL | 85.4 (34.1) | 89.4 (127.1)
Statistical Analysis 1: Comparison: Part 2: Atezolizumab IV 1200 mg vs Part 2: Atezolizumab SC 1875 mg; Test type: Non-Inferiority — The null hypothesis that atezolizumab SC is inferior to atezolizumab IV is rejected if the lower bound of the 2-sided 90% confidence interval [CI] of the geometric mean ratio is greater than or equal to (≥) the non-inferiority margin 0.8; Geometric mean ratio = 1.05, 90.0% CI 2-sided [0.88 to 1.24]

3. Primary Outcome: Part 2: Area Under the Concentration-Time Curve From Time Zero to 21 Days (AUC 0-21 d) at Cycle 1
Time Frame: From start of dosing up to Day 21 in Cycle 1 (Cycle length = 21 days)
Population: PK-evaluable population included all participants who received at least one dose of atezolizumab and had at least 1 evaluable post dose PK sample that could affect PK results. Overall number analyzed is the number of participants with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms day per mL (μg*day/mL)
Arm/Group | Part 2: Atezolizumab IV 1200 mg | Part 2: Atezolizumab SC 1875 mg
Number analyzed (Participants) | 122 | 246
micrograms day per mL (μg*day/mL) | 3327.9 (19.4) | 2907.1 (35.9)
Statistical Analysis 1: Comparison: Part 2: Atezolizumab IV 1200 mg vs Part 2: Atezolizumab SC 1875 mg; Test type: Non-Inferiority — The null hypothesis that atezolizumab SC is inferior to atezolizumab IV is rejected if the lower bound of the 2-sided 90% CI of the geometric mean ratio is ≥ the non-inferiority margin 0.8; Geometric mean ratio = 0.87, 90.0% CI 2-sided [0.83 to 0.92]

4. Secondary Outcome: Part 1: Maximum Observed Serum Concentration (Cmax) of Atezolizumab
Time Frame: Predose and post dose on Day 1 of Cycle 1 and post dose on Days 3 and 8 of Cycle 1 (Cycle length = 21 days for cohorts 1 and 3 and 14 days for cohort 2)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 1 Cohort 1: Atezolizumab SC Co-mix 1800 mg | Part 1 Cohort 2: Atezolizumab SC Co-mix 1200 mg | Part 1 Cohort 3: Atezolizumab SC Co-mix 1800 mg
Number analyzed (Participants) | 13 | 14 | 30
μg/mL | 251 (40.9) | 129 (42.5) | 181 (38.3)

5. Secondary Outcome: Part 1: Time to Maximum Serum Concentration (Tmax) of Atezolizumab
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Median (Full Range); unit: days
Arm/Group | Part 1 Cohort 1: Atezolizumab SC Co-mix 1800 mg | Part 1 Cohort 2: Atezolizumab SC Co-mix 1200 mg | Part 1 Cohort 3: Atezolizumab SC Co-mix 1800 mg
Number analyzed (Participants) | 13 | 14 | 30
days | 3.02 [2.93 to 7.80] | 3.45 [3.00 to 8.95] | 3.92 [2.99 to 7.11]

6. Secondary Outcome: Part 1: Area Under the Concentration-time Curve (AUClast) of Atezolizumab
Time Frame: Predose and up to 21 days post dose in Cycle 1 for cohorts 1 and 3 and from predose up to 14 days post last dose in Cycle 1 for cohort 2 (Cycle length= 21 days for cohorts 1 and 3 and 14 days for cohort 2)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*day/mL
Arm/Group | Part 1 Cohort 1: Atezolizumab SC Co-mix 1800 mg | Part 1 Cohort 2: Atezolizumab SC Co-mix 1200 mg | Part 1 Cohort 3: Atezolizumab SC Co-mix 1800 mg
Number analyzed (Participants) | 13 | 14 | 30
μg*day/mL | 3870 (38.6) | 1410 (41.8) | 2820 (38.6)

7. Secondary Outcome: Part 1: Serum Atezolizumab Concentration at Specified Timepoint During SC Administration
Description: Cycle length =21 days for cohorts 1 and 3 and 14 days for cohort 2. Day=D; Cycle=C.
Time Frame: Cohort 1: Predose: D1 & postdose: D1, 3, 8 of C1; Cohort 2: Pre & postdose: D1 of C1, 3 & postdose: D3, 8 of C1, Predose: D1 of C2; Cohort 3: Pre & postdose: D1 of C1, 2 & postdose: D3, 8 of C1, D2, 4 & 9 of C2 & pre dose: D1 of C3
Population: PK-evaluable population included all participants who received at least one dose of atezolizumab and had at least 1 evaluable post dose PK sample that could affect PK results. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at a given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 1 Cohort 1: Atezolizumab SC Co-mix 1800 mg | Part 1 Cohort 2: Atezolizumab SC Co-mix 1200 mg | Part 1 Cohort 3: Atezolizumab SC Co-mix 1800 mg
Number analyzed (Participants) | 13 | 15 | 39
μg/mL
  Cycle 1, Day 1: Pre-dose | NA (NA) — The data was not evaluable as all the samples were below lower limit of quantification (BLLQ). | NA (NA) — The data was not evaluable as all the samples were BLLQ. | NA (NA) — The data was not evaluable as all the samples were BLLQ.
  Cycle 1, Day 1: Post-dose | 116 (57.8) | 61.7 (70.9) | 108 (57.6)
  Cycle 1, Day 3: Post-dose: number analyzed (Participants) | 13 | 15 | 38
  Cycle 1, Day 3: Post-dose | 247 (40.5) | 123 (44.3) | 166 (45.7)
  Cycle 1, Day 8: Post-dose: number analyzed (Participants) | 13 | 15 | 37
  Cycle 1, Day 8: Post-dose | 230 (36.6) | 110 (45.0) | 162 (43.5)
  Cycle 2, Day 1: Pre-dose: number analyzed (Participants) | 0 | 15 | 35
  Cycle 2, Day 1: Pre-dose |  | 77.5 (51.4) | 78.3 (88.6)
  Cycle 2, Day 1: Post-dose: number analyzed (Participants) | 0 | 0 | 36
  Cycle 2, Day 1: Post-dose |  |  | 87.7 (64.7)
  Cycle 2, Day 2: Post-dose: number analyzed (Participants) | 0 | 0 | 36
  Cycle 2, Day 2: Post-dose |  |  | 183 (46.1)
  Cycle 2, Day 4: Post-dose: number analyzed (Participants) | 0 | 0 | 34
  Cycle 2, Day 4: Post-dose |  |  | 245 (42.0)
  Cycle 2, Day 9: Post-dose: number analyzed (Participants) | 0 | 0 | 35
  Cycle 2, Day 9: Post-dose |  |  | 225 (37.2)
  Cycle 3, Day 1: Pre-dose: number analyzed (Participants) | 0 | 14 | 33
  Cycle 3, Day 1: Pre-dose |  | 104 (47.8) | 123 (57.2)
  Cycle 3, Day 1: Post-dose: number analyzed (Participants) | 0 | 1 | 0
  Cycle 3, Day 1: Post-dose |  | 189 (NA) — Since only 1 participant was analysed the geometric coefficient of variation could not be calculated. |

8. Secondary Outcome: Part 1: Percentage of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as AEs. AEs were reported based on the National Cancer Institute Common Terminology Criteria for AEs, version 5.0 (NCI-CTCAE, v5.0). Percentages have been rounded to one decimal place.
Time Frame: From initiation of study treatment up to approximately 69 months
Population: Safety-evaluable population included all participants who received at least one dose of atezolizumab (IV or SC), with participants grouped according to treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohort 1: Atezolizumab SC Co-mix 1800 mg | Part 1 Cohort 2: Atezolizumab SC Co-mix 1200 mg | Part 1 Cohort 3: Atezolizumab SC Co-mix 1800 mg
Number analyzed (Participants) | 13 | 15 | 39
percentage of participants | 100 | 86.7 | 84.6

9. Secondary Outcome: Part 2: Percentage of Participants With AEs
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as AEs. AEs were reported based on the NCI-CTCAE, V5.0. Percentages have been rounded to one decimal place.
Time Frame: From initiation of study treatment up to approximately 44.7 months
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Atezolizumab IV 1200 mg | Part 2: Atezolizumab SC 1875 mg
Number analyzed (Participants) | 124 | 247
percentage of participants | 85.5 | 89.9

10. Secondary Outcome: Part 2: Model Predicted Ctrough of Atezolizumab at Cycle 1
Time Frame: Cycle 1 (Cycle length=21 days)
Population: PK evaluable population included all participants randomized to the atezolizumab SC and atezolizumab IV treatment arms with at least one post-baseline PK sample. Overall number analyzed is the number of participants with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 2: Atezolizumab IV 1200 mg | Part 2: Atezolizumab SC 1875 mg
Number analyzed (Participants) | 122 | 246
μg/mL | 88.7 (26.2) | 97.2 (42.3)

11. Secondary Outcome: Part 2: Model Predicted Ctrough at Steady State (Ctrough,ss) of Atezolizumab
Description: 1 cycle=21 days Abbreviations used-Cycle=C; Day =D; Atezolizumab=atezo.
Time Frame: Atezo SC: Pre&postdose C1D1, postdose C1 Days 2,4,8, Pre&postdose C2,D1 and Predose on D1 of C3,4,8,12 and 16 ; Atezo IV: Pre&postdose on C1D1, postdose C1 Days 2,4,8; Pre&postdose C2D1, Predose on D1 of C3,4,8,12, and 16 (up to approximately 16 months)
Population: PK-evaluable population included all participants who received at least one dose of atezolizumab (atezolizumab SC or atezolizumab IV) and had at least 1 evaluable post dose PK sample. Overall number analyzed is the number of participants with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 2: Atezolizumab IV 1200 mg | Part 2: Atezolizumab SC 1875 mg
Number analyzed (Participants) | 122 | 246
μg/mL | 179 (38.8) | 205 (58.1)

12. Secondary Outcome: Part 2: Model Predicted AUC at Steady State (AUCss) of Atezolizumab
Description: 1 cycle=21 days Abbreviations used-Cycle=C; Day =D; Atezolizumab=atezo
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*day/mL
Arm/Group | Part 2: Atezolizumab IV 1200 mg | Part 2: Atezolizumab SC 1875 mg
Number analyzed (Participants) | 122 | 246
ug*day/mL | 6107 (27.3) | 6163 (46.7)

13. Secondary Outcome: Part 2: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants having a complete response (CR) or partial response (PR) as determined by investigator assessment of radiographic disease per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST V1.1). CR was defined as the disappearance of all target lesions and any pathological lymph nodes must have reduction in short axis to < 10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters (SOD) of all target lesions, taking as reference the baseline SOD in the absence of CR. Percentage of participants who achieved confirmed objective response (CR or PR) have been reported. Percentages have been rounded to one decimal place.
Time Frame: Up to approximately 25 months
Population: Response-evaluable population included all participants with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: Atezolizumab IV 1200 mg | Part 2: Atezolizumab SC 1875 mg
Number analyzed (Participants) | 124 | 245
percentage of participants | 10.5 [5.7 to 17.3] | 11.0 [7.4 to 15.6]
Statistical Analysis 1: Comparison: Part 2: Atezolizumab IV 1200 mg vs Part 2: Atezolizumab SC 1875 mg; Test type: Superiority; p = 0.8757, Cochran-Mantel-Haenszel; Difference in ORR = 0.54, 95% CI 2-sided [-6.56 to 7.63]

14. Secondary Outcome: Part 2: Progression-free Survival (PFS)
Description: PFS was defined as the time from study start to the first occurrence of PD, as determined by the investigator according to RECIST v1.1 or death from any cause (whichever occurs first). PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest SOD at prior timepoints (including baseline). In addition to the relative increase of 20%, the SOD must also demonstrate an absolute increase of ≥ 5 mm. PFS was analyzed using the Kaplan-Meier method.
Time Frame: Up to approximately 25 months
Population: FAS included all randomized participants, with participants grouped according to their assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: Atezolizumab IV 1200 mg | Part 2: Atezolizumab SC 1875 mg
Number analyzed (Participants) | 124 | 247
months | 2.9 [1.8 to 4.2] | 2.8 [2.7 to 4.1]
Statistical Analysis 1: Comparison: Part 2: Atezolizumab IV 1200 mg vs Part 2: Atezolizumab SC 1875 mg; Test type: Superiority; p = 0.6906, Log Rank; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.83 to 1.33]

15. Secondary Outcome: Part 2: Overall Survival (OS)
Description: OS was defined as the time from the date of study randomization to the date of death from any cause.
Time Frame: Up to approximately 44.7 months
Population: FAS included all randomized participants, with participants grouped according to their assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: Atezolizumab IV 1200 mg | Part 2: Atezolizumab SC 1875 mg
Number analyzed (Participants) | 124 | 247
months | 10.1 [7.5 to 12.3] | 10.9 [8.5 to 14.4]
Statistical Analysis 1: Comparison: Part 2: Atezolizumab IV 1200 mg vs Part 2: Atezolizumab SC 1875 mg; Test type: Superiority; p = 0.9766, Log Rank; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.78 to 1.27]

16. Secondary Outcome: Part 2: Duration of Response (DOR)
Description: DOR was defined as the time from first occurrence of a documented confirmed objective response (CR or PR) to PD as determined by the investigator according to RECIST v1.1. or death from any cause, whichever occurs first. CR was defined as the disappearance of all target lesions and any pathological lymph nodes must have a reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD in the absence of CR. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest SOD at prior timepoints (including baseline). In addition to the relative increase of 20%, the SODs must also demonstrate an absolute increase of ≥ 5 mm.
Time Frame: Up to approximately 25 months
Population: DOR-evaluable population included all participants with a measurable disease at baseline and a post-baseline confirmed objective response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: Atezolizumab IV 1200 mg | Part 2: Atezolizumab SC 1875 mg
Number analyzed (Participants) | 13 | 27
months | 11.2 [4.2 to NA] — The upper limit of the 95% confidence interval (CI) was not estimable due to an insufficient number of participants with events. | 15.1 [5.6 to NA] — The upper limit of the 95% CI was not estimable due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: Part 2: Atezolizumab IV 1200 mg vs Part 2: Atezolizumab SC 1875 mg; Test type: Superiority; p = 0.8375, Log Rank; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.34 to 2.42]

17. Secondary Outcome: Part 2: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Item Library (IL) 57 Physical Functioning Score
Description: EORTC IL57 questionnaire has 10 items and covers 3 scales: physical functioning (PF), role functioning (RF) & global health status/quality of life (GHS/QoL) & 1 item from EORTC IL. PF scale has 5 items evaluating the extent to which participants have trouble doing strenuous activities; taking long walks & short walks; need to stay in bed or a chair; need help with eating, dressing, bathing/using toilet. RF scale has 2 items evaluating extent to which participants are limited in doing work & pursuing leisure activities in previous week. GHS/QoL scale has 2 items evaluating participants' overall health & QoL in previous week. Questions are answered on a 4-point Likert scale (where 1="Not at all" to 4="Very much") for physical and role functioning & a 7-point scale (where 1="Very poor" to 7="Excellent") for GHS/QoL. For each scale, mean of the items are linearly transformed to obtain scores from 0-100, where 100 = best possible score. Higher score indicates better outcome.
Time Frame: Baseline, Day 1 of Cycles 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 34, 36, 38, 40, 42, 44, 46, 48, 50, 52, 54, 56, 58, 60, 62, 64 (Cycle length = 21 days), and Treatment Discontinuation Visit (up to approximately 44 months)
Population: FAS included all randomized participants, with participants grouped according to their assigned treatment. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 2: Atezolizumab IV 1200 mg | Part 2: Atezolizumab SC 1875 mg
Number analyzed (Participants) | 117 | 243
score on a scale
  Baseline | 74.53 (20.37) | 72.15 (21.94)
  Change at Day 1 Cycle 2: number analyzed (Participants) | 106 | 219
  Change at Day 1 Cycle 2 | -6.23 (19.17) | -4.23 (17.01)
  Change at Day 1 Cycle 3: number analyzed (Participants) | 86 | 183
  Change at Day 1 Cycle 3 | -4.55 (19.04) | -4.99 (17.63)
  Change at Day 1 Cycle 4: number analyzed (Participants) | 80 | 167
  Change at Day 1 Cycle 4 | -5.75 (22.04) | -4.47 (20.86)
  Change at Day 1 Cycle 5: number analyzed (Participants) | 64 | 134
  Change at Day 1 Cycle 5 | -1.46 (21.40) | -2.14 (20.05)
  Change at Day 1 Cycle 6: number analyzed (Participants) | 58 | 120
  Change at Day 1 Cycle 6 | -2.76 (25.68) | -0.67 (20.09)
  Change at Day 1 Cycle 8: number analyzed (Participants) | 47 | 95
  Change at Day 1 Cycle 8 | -0.14 (19.24) | -0.42 (19.76)
  Change at Day 1 Cycle 10: number analyzed (Participants) | 41 | 81
  Change at Day 1 Cycle 10 | -1.46 (22.39) | 0.82 (20.96)
  Change at Day 1 Cycle 12: number analyzed (Participants) | 35 | 70
  Change at Day 1 Cycle 12 | 0.95 (22.64) | 1.14 (20.43)
  Change at Day 1 Cycle 14: number analyzed (Participants) | 30 | 60
  Change at Day 1 Cycle 14 | 0.67 (19.37) | 1.11 (18.82)
  Change at Day 1 Cycle 16: number analyzed (Participants) | 28 | 53
  Change at Day 1 Cycle 16 | -2.14 (23.38) | 2.26 (19.30)
  Change at Day 1 Cycle 18: number analyzed (Participants) | 23 | 50
  Change at Day 1 Cycle 18 | -0.87 (19.10) | 0.67 (19.30)
  Change at Day 1 Cycle 20: number analyzed (Participants) | 21 | 44
  Change at Day 1 Cycle 20 | -1.59 (22.30) | -0.15 (19.53)
  Change at Day 1 Cycle 22: number analyzed (Participants) | 18 | 36
  Change at Day 1 Cycle 22 | -2.22 (23.54) | -1.67 (23.66)
  Change at Day 1 Cycle 24: number analyzed (Participants) | 16 | 34
  Change at Day 1 Cycle 24 | -0.83 (22.69) | -1.76 (20.97)
  Change at Day 1 Cycle 26: number analyzed (Participants) | 16 | 31
  Change at Day 1 Cycle 26 | 0.83 (17.36) | -1.94 (23.61)
  Change at Day 1 Cycle 28: number analyzed (Participants) | 14 | 23
  Change at Day 1 Cycle 28 | 2.38 (14.70) | 0.51 (19.46)
  Change at Day 1 Cycle 30: number analyzed (Participants) | 13 | 21
  Change at Day 1 Cycle 30 | 2.05 (16.42) | 0.95 (18.89)
  Change at Day 1 Cycle 32: number analyzed (Participants) | 12 | 22
  Change at Day 1 Cycle 32 | -6.67 (21.27) | 0.61 (22.34)
  Change at Day 1 Cycle 34: number analyzed (Participants) | 11 | 20
  Change at Day 1 Cycle 34 | -2.42 (16.40) | 3.00 (26.62)
  Change at Day 1 Cycle 36: number analyzed (Participants) | 11 | 20
  Change at Day 1 Cycle 36 | 0.61 (17.24) | 6.00 (23.59)
  Change at Day 1 Cycle 38: number analyzed (Participants) | 11 | 18
  Change at Day 1 Cycle 38 | 3.64 (17.22) | 4.07 (24.96)
  Change at Day 1 Cycle 40: number analyzed (Participants) | 11 | 18
  Change at Day 1 Cycle 40 | 0.00 (25.65) | 1.11 (23.79)
  Change at Day 1 Cycle 42: number analyzed (Participants) | 8 | 18
  Change at Day 1 Cycle 42 | 1.67 (19.76) | 2.96 (21.36)
  Change at Day 1 Cycle 44: number analyzed (Participants) | 8 | 16
  Change at Day 1 Cycle 44 | 5.83 (12.57) | 5.00 (21.15)
  Change at Day 1 Cycle 46: number analyzed (Participants) | 8 | 17
  Change at Day 1 Cycle 46 | 5.83 (16.88) | 5.88 (26.34)
  Change at Day 1 Cycle 48: number analyzed (Participants) | 7 | 14
  Change at Day 1 Cycle 48 | 8.57 (10.69) | 8.10 (24.13)
  Change at Day 1 Cycle 50: number analyzed (Participants) | 7 | 11
  Change at Day 1 Cycle 50 | 4.76 (14.76) | 9.09 (29.25)
  Change at Day 1 Cycle 52: number analyzed (Participants) | 6 | 10
  Change at Day 1 Cycle 52 | 12.22 (12.94) | 5.33 (24.30)
  Change at Day 1 Cycle 54: number analyzed (Participants) | 3 | 8
  Change at Day 1 Cycle 54 | 11.11 (10.18) | 6.67 (29.81)
  Change at Day 1 Cycle 56: number analyzed (Participants) | 2 | 3
  Change at Day 1 Cycle 56 | 10.00 (4.71) | 8.89 (13.88)
  Change at Day 1 Cycle 58: number analyzed (Participants) | 1 | 2
  Change at Day 1 Cycle 58 | 6.67 (NA) — Standard deviation (SD) was not estimable since only 1 participant was evaluated. | 3.33 (14.14)
  Change at Day 1 Cycle 60: number analyzed (Participants) | 1 | 1
  Change at Day 1 Cycle 60 | 20.00 (NA) — SD was not estimable since only 1 participant was evaluated. | 13.33 (NA) — SD was not estimable since only 1 participant was evaluated.
  Change at Day 1 Cycle 62: number analyzed (Participants) | 1 | 1
  Change at Day 1 Cycle 62 | 13.33 (NA) — SD was not estimable since only 1 participant was evaluated. | 13.33 (NA) — SD was not estimable since only 1 participant was evaluated.
  Change at Day 1 Cycle 64: number analyzed (Participants) | 0 | 1
  Change at Day 1 Cycle 64 |  | 13.33 (NA) — SD was not estimable since only 1 participant was evaluated.
  Change at Treatment Discontinuation Visit: number analyzed (Participants) | 74 | 149
  Change at Treatment Discontinuation Visit | -19.01 (28.26) | -15.68 (25.67)

18. Secondary Outcome: Part 2: Change From Baseline in EORTC IL57 Role Functioning Score
Description: EORTC IL57 questionnaire has 10 items and covers 3 scales: PF, RF & GHS/QoL & 1 item from EORTC IL. PF scale has 5 items evaluating the extent to which participants have trouble doing strenuous activities; taking long walks & short walks; need to stay in bed or a chair; need help with eating, dressing, bathing/using toilet. RF scale has 2 items evaluating extent to which participants are limited in doing work & pursuing leisure activities in previous week. GHS/QoL scale has 2 items evaluating participants' overall health & QoL in previous week. Questions are answered on a 4-point Likert scale (where 1="Not at all" to 4="Very much") for physical and role functioning & a 7-point scale (where 1="Very poor" to 7="Excellent") for GHS/QoL. For each scale, mean of the items are linearly transformed to obtain scores from 0-100, where 100 = best possible score. Higher score indicates better outcome.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 2: Atezolizumab IV 1200 mg | Part 2: Atezolizumab SC 1875 mg
Number analyzed (Participants) | 117 | 242
score on a scale
  Baseline | 74.93 (25.67) | 74.86 (27.51)
  Change at Day 1 Cycle 2: number analyzed (Participants) | 106 | 218
  Change at Day 1 Cycle 2 | 0.31 (29.46) | -4.36 (24.48)
  Change at Day 1 Cycle 3: number analyzed (Participants) | 86 | 182
  Change at Day 1 Cycle 3 | -3.29 (27.51) | -4.67 (25.83)
  Change at Day 1 Cycle 4: number analyzed (Participants) | 80 | 167
  Change at Day 1 Cycle 4 | -0.83 (26.90) | -6.59 (28.63)
  Change at Day 1 Cycle 5: number analyzed (Participants) | 64 | 134
  Change at Day 1 Cycle 5 | 2.34 (31.13) | -5.22 (30.27)
  Change at Day 1 Cycle 6: number analyzed (Participants) | 58 | 119
  Change at Day 1 Cycle 6 | 0.00 (32.14) | -5.74 (29.39)
  Change at Day 1 Cycle 8: number analyzed (Participants) | 47 | 94
  Change at Day 1 Cycle 8 | 4.96 (29.47) | -1.95 (25.50)
  Change at Day 1 Cycle 10: number analyzed (Participants) | 41 | 81
  Change at Day 1 Cycle 10 | 1.63 (29.06) | -0.82 (24.71)
  Change at Day 1 Cycle 12: number analyzed (Participants) | 35 | 69
  Change at Day 1 Cycle 12 | 4.29 (29.80) | -2.66 (30.20)
  Change at Day 1 Cycle 14: number analyzed (Participants) | 30 | 60
  Change at Day 1 Cycle 14 | 6.11 (22.09) | -3.61 (30.24)
  Change at Day 1 Cycle 16: number analyzed (Participants) | 28 | 53
  Change at Day 1 Cycle 16 | -0.60 (29.91) | -1.26 (27.12)
  Change at Day 1 Cycle 18: number analyzed (Participants) | 23 | 50
  Change at Day 1 Cycle 18 | 0.72 (21.60) | -2.00 (27.90)
  Change at Day 1 Cycle 20: number analyzed (Participants) | 21 | 44
  Change at Day 1 Cycle 20 | 7.94 (30.10) | -2.65 (27.83)
  Change at Day 1 Cycle 22: number analyzed (Participants) | 18 | 36
  Change at Day 1 Cycle 22 | 6.48 (28.66) | -5.09 (34.23)
  Change at Day 1 Cycle 24: number analyzed (Participants) | 16 | 34
  Change at Day 1 Cycle 24 | 3.13 (24.51) | -4.41 (29.39)
  Change at Day 1 Cycle 26: number analyzed (Participants) | 16 | 31
  Change at Day 1 Cycle 26 | 4.17 (36.77) | 0.54 (27.38)
  Change at Day 1 Cycle 28: number analyzed (Participants) | 14 | 23
  Change at Day 1 Cycle 28 | 7.14 (16.94) | 5.07 (29.91)
  Change at Day 1 Cycle 30: number analyzed (Participants) | 13 | 21
  Change at Day 1 Cycle 30 | -2.56 (20.24) | 3.17 (31.01)
  Change at Day 1 Cycle 32: number analyzed (Participants) | 12 | 22
  Change at Day 1 Cycle 32 | -6.94 (19.41) | -0.76 (31.49)
  Change at Day 1 Cycle 34: number analyzed (Participants) | 11 | 20
  Change at Day 1 Cycle 34 | -6.06 (22.70) | 0.00 (34.20)
  Change at Day 1 Cycle 36: number analyzed (Participants) | 11 | 20
  Change at Day 1 Cycle 36 | -3.03 (17.98) | 1.67 (31.48)
  Change at Day 1 Cycle 38: number analyzed (Participants) | 11 | 18
  Change at Day 1 Cycle 38 | 4.55 (16.82) | 5.56 (26.20)
  Change at Day 1 Cycle 40: number analyzed (Participants) | 11 | 18
  Change at Day 1 Cycle 40 | 1.52 (24.10) | 1.85 (28.52)
  Change at Day 1 Cycle 42: number analyzed (Participants) | 8 | 18
  Change at Day 1 Cycle 42 | -6.25 (23.46) | 3.70 (32.11)
  Change at Day 1 Cycle 44: number analyzed (Participants) | 8 | 16
  Change at Day 1 Cycle 44 | -2.08 (16.52) | 7.29 (31.60)
  Change at Day 1 Cycle 46: number analyzed (Participants) | 8 | 17
  Change at Day 1 Cycle 46 | 0.00 (23.57) | 4.90 (32.68)
  Change at Day 1 Cycle 48: number analyzed (Participants) | 7 | 14
  Change at Day 1 Cycle 48 | 2.38 (20.25) | 8.33 (31.86)
  Change at Day 1 Cycle 50: number analyzed (Participants) | 7 | 11
  Change at Day 1 Cycle 50 | 2.38 (20.25) | 13.64 (36.38)
  Change at Day 1 Cycle 52: number analyzed (Participants) | 6 | 10
  Change at Day 1 Cycle 52 | 2.78 (28.71) | 1.67 (24.15)
  Change at Day 1 Cycle 54: number analyzed (Participants) | 3 | 8
  Change at Day 1 Cycle 54 | -11.11 (34.69) | 2.08 (36.12)
  Change at Day 1 Cycle 56: number analyzed (Participants) | 2 | 3
  Change at Day 1 Cycle 56 | 0.00 (23.57) | -5.56 (19.25)
  Change at Day 1 Cycle 58: number analyzed (Participants) | 1 | 2
  Change at Day 1 Cycle 58 | -33.33 (NA) — SD was not estimable since only 1 participant was evaluated. | 0.00 (23.57)
  Change at Day 1 Cycle 60: number analyzed (Participants) | 1 | 1
  Change at Day 1 Cycle 60 | 16.67 (NA) — SD was not estimable since only 1 participant was evaluated. | 16.67 (NA) — SD was not estimable since only 1 participant was evaluated.
  Change at Day 1 Cycle 62: number analyzed (Participants) | 1 | 1
  Change at Day 1 Cycle 62 | 16.67 (NA) — SD was not estimable since only 1 participant was evaluated. | 16.67 (NA) — SD was not estimable since only 1 participant was evaluated.
  Change at Day 1 Cycle 64: number analyzed (Participants) | 0 | 1
  Change at Day 1 Cycle 64 |  | 16.67 (NA) — SD was not estimable since only 1 participant was evaluated.
  Change at Treatment Discontinuation Visit: number analyzed (Participants) | 74 | 149
  Change at Treatment Discontinuation Visit | -20.27 (33.70) | -21.14 (34.80)

19. Secondary Outcome: Part 2: Change From Baseline in EORTC IL57 Global Health Status Score
Description: as for outcome 18
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 2: Atezolizumab IV 1200 mg | Part 2: Atezolizumab SC 1875 mg
Number analyzed (Participants) | 117 | 242
score on a scale
  Baseline | 66.52 (17.68) | 63.50 (22.00)
  Change at Day 1 Cycle 2: number analyzed (Participants) | 106 | 218
  Change at Day 1 Cycle 2 | -3.54 (21.33) | -2.48 (21.77)
  Change at Day 1 Cycle 3: number analyzed (Participants) | 86 | 182
  Change at Day 1 Cycle 3 | -2.91 (20.92) | -1.83 (23.04)
  Change at Day 1 Cycle 4: number analyzed (Participants) | 80 | 167
  Change at Day 1 Cycle 4 | -2.71 (19.61) | -2.25 (22.21)
  Change at Day 1 Cycle 5: number analyzed (Participants) | 64 | 134
  Change at Day 1 Cycle 5 | 0.65 (19.26) | -1.43 (25.35)
  Change at Day 1 Cycle 6: number analyzed (Participants) | 58 | 119
  Change at Day 1 Cycle 6 | -0.14 (21.99) | 0.14 (22.94)
  Change at Day 1 Cycle 8: number analyzed (Participants) | 47 | 94
  Change at Day 1 Cycle 8 | 3.01 (18.26) | 1.86 (22.74)
  Change at Day 1 Cycle 10: number analyzed (Participants) | 41 | 81
  Change at Day 1 Cycle 10 | 5.28 (19.87) | 0.72 (23.17)
  Change at Day 1 Cycle 12: number analyzed (Participants) | 35 | 69
  Change at Day 1 Cycle 12 | 6.19 (18.45) | -2.78 (18.56)
  Change at Day 1 Cycle 14: number analyzed (Participants) | 30 | 60
  Change at Day 1 Cycle 14 | 7.50 (17.42) | 1.94 (19.67)
  Change at Day 1 Cycle 16: number analyzed (Participants) | 28 | 53
  Change at Day 1 Cycle 16 | 6.55 (17.77) | 1.73 (18.52)
  Change at Day 1 Cycle 18: number analyzed (Participants) | 23 | 50
  Change at Day 1 Cycle 18 | 4.71 (19.11) | 0.67 (17.56)
  Change at Day 1 Cycle 20: number analyzed (Participants) | 21 | 44
  Change at Day 1 Cycle 20 | 9.52 (16.73) | -0.95 (18.52)
  Change at Day 1 Cycle 22: number analyzed (Participants) | 18 | 36
  Change at Day 1 Cycle 22 | 5.56 (21.20) | 0.00 (19.92)
  Change at Day 1 Cycle 24: number analyzed (Participants) | 16 | 34
  Change at Day 1 Cycle 24 | 7.29 (28.20) | -2.70 (18.99)
  Change at Day 1 Cycle 26: number analyzed (Participants) | 16 | 31
  Change at Day 1 Cycle 26 | 1.56 (24.95) | -2.15 (21.51)
  Change at Day 1 Cycle 28: number analyzed (Participants) | 14 | 23
  Change at Day 1 Cycle 28 | 1.79 (16.72) | 1.81 (21.17)
  Change at Day 1 Cycle 30: number analyzed (Participants) | 13 | 21
  Change at Day 1 Cycle 30 | 5.77 (16.45) | 3.17 (21.81)
  Change at Day 1 Cycle 32: number analyzed (Participants) | 12 | 22
  Change at Day 1 Cycle 32 | 0.00 (18.46) | 0.38 (17.91)
  Change at Day 1 Cycle 34: number analyzed (Participants) | 11 | 20
  Change at Day 1 Cycle 34 | 0.00 (20.07) | 2.50 (19.70)
  Change at Day 1 Cycle 36: number analyzed (Participants) | 11 | 20
  Change at Day 1 Cycle 36 | -1.52 (15.73) | 1.67 (20.52)
  Change at Day 1 Cycle 38: number analyzed (Participants) | 11 | 18
  Change at Day 1 Cycle 38 | 2.27 (21.11) | 3.70 (20.66)
  Change at Day 1 Cycle 40: number analyzed (Participants) | 11 | 18
  Change at Day 1 Cycle 40 | 5.30 (21.50) | 1.39 (19.85)
  Change at Day 1 Cycle 42: number analyzed (Participants) | 8 | 18
  Change at Day 1 Cycle 42 | 0.00 (17.25) | 2.31 (20.37)
  Change at Day 1 Cycle 44: number analyzed (Participants) | 8 | 16
  Change at Day 1 Cycle 44 | 2.08 (18.23) | 3.65 (19.95)
  Change at Day 1 Cycle 46: number analyzed (Participants) | 8 | 17
  Change at Day 1 Cycle 46 | 2.08 (25.88) | 2.45 (21.60)
  Change at Day 1 Cycle 48: number analyzed (Participants) | 7 | 14
  Change at Day 1 Cycle 48 | 7.14 (15.54) | 4.17 (20.35)
  Change at Day 1 Cycle 50: number analyzed (Participants) | 7 | 11
  Change at Day 1 Cycle 50 | -2.38 (17.16) | 3.03 (21.82)
  Change at Day 1 Cycle 52: number analyzed (Participants) | 6 | 10
  Change at Day 1 Cycle 52 | 8.33 (12.91) | -3.33 (16.76)
  Change at Day 1 Cycle 54: number analyzed (Participants) | 3 | 8
  Change at Day 1 Cycle 54 | -2.78 (12.73) | 0.00 (22.27)
  Change at Day 1 Cycle 56: number analyzed (Participants) | 2 | 3
  Change at Day 1 Cycle 56 | 4.17 (5.89) | 2.78 (4.81)
  Change at Day 1 Cycle 58: number analyzed (Participants) | 1 | 2
  Change at Day 1 Cycle 58 | 0.00 (NA) — SD was not estimable since only 1 participant was evaluated. | 0.00 (0.00)
  Change at Day 1 Cycle 60: number analyzed (Participants) | 1 | 1
  Change at Day 1 Cycle 60 | 8.33 (NA) — SD was not estimable since only 1 participant was evaluated. | 0.00 (NA) — SD was not estimable since only 1 participant was evaluated.
  Change at Day 1 Cycle 62: number analyzed (Participants) | 1 | 1
  Change at Day 1 Cycle 62 | -8.33 (NA) — SD was not estimable since only 1 participant was evaluated. | 0.00 (NA) — SD was not estimable since only 1 participant was evaluated.
  Change at Day 1 Cycle 64: number analyzed (Participants) | 0 | 1
  Change at Day 1 Cycle 64 |  | 0.00 (NA) — SD was not estimable since only 1 participant was evaluated.
  Change at Treatment Discontinuation Visit: number analyzed (Participants) | 74 | 149
  Change at Treatment Discontinuation Visit | -14.53 (26.28) | -13.37 (25.42)

20. Secondary Outcome: Part 2: Overall Satisfaction With Treatment Over Time, Assessed by the Modified Satisfaction With Therapy (SWT) Scale of the Cancer Therapy Satisfaction Questionnaire (CTSQ)
Description: Modified SWT scale of the CTSQ consisted of seven items that measured seven domains related to satisfaction with cancer therapy. These include worthwhile, difficulty, benefits, feelings about side effects, form of therapy, overall satisfaction, and if participants would choose the therapy taking everything into consideration. Each domain is rated on a 5-point scale, with 1 representing the worst response and 5 representing the best response, except in the case of one reverse-scored item. Mean of the items were linearly transformed to obtain scores from 0-100, where 100 was the best possible score. Higher scores indicate higher satisfaction. Here, data for 'overall satisfaction' domain has been presented.
Time Frame: Day 1 Cycle 3 or Treatment Discontinuation Visit (if treatment discontinued at any visit before Cycle 3) (Cycle length = 21 days)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 2: Atezolizumab IV 1200 mg | Part 2: Atezolizumab SC 1875 mg
Number analyzed (Participants) | 98 | 191
score on a scale
  Day 1 Cycle 3: number analyzed (Participants) | 83 | 162
  Day 1 Cycle 3 | 77.29 (16.08) | 75.56 (18.61)
  Treatment Discontinuation Visit: number analyzed (Participants) | 15 | 29
  Treatment Discontinuation Visit | 50.67 (19.90) | 61.21 (19.81)

21. Secondary Outcome: Part 2: Percentage of Participants by Their Responses to AE's Burden Over Time, Assessed by the Treatment-related Symptom Burden Item From the EORTC IL57
Description: The overall patient-reported AE burden was assessed using a single item from the EORTC IL57 questionnaire i.e "To what extent have you been troubled with side-effects from your treatment?" The questions were answered on a 4-point Likert scale, where 1="Not at all" to 4="Very much". Higher scores indicated greater AE burden. Percentages have been rounded to one decimal place.
Time Frame: Baseline, Day 1 of Cycles 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 34, 36, 38, 40, 42, 44, 46, 48, 50, 52, 54, 56, 58, 60, 62, and 64 (Cycle length = 21 days)
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Atezolizumab IV 1200 mg | Part 2: Atezolizumab SC 1875 mg
Number analyzed (Participants) | 113 | 238
percentage of participants
  Baseline - Not at all | 49.6 | 56.7
  Baseline - A little | 36.3 | 28.6
  Baseline - Quite a bit | 8.0 | 10.1
  Baseline - Very much | 6.2 | 4.6
  Day 1 Cycle 2 - Not at all: number analyzed (Participants) | 108 | 222
  Day 1 Cycle 2 - Not at all | 47.2 | 49.5
  Day 1 Cycle 2 - A little: number analyzed (Participants) | 108 | 222
  Day 1 Cycle 2 - A little | 39.8 | 35.6
  Day 1 Cycle 2 - Quite a bit: number analyzed (Participants) | 108 | 222
  Day 1 Cycle 2 - Quite a bit | 9.3 | 12.6
  Day 1 Cycle 2 - Very much: number analyzed (Participants) | 108 | 222
  Day 1 Cycle 2 - Very much | 3.7 | 2.3
  Day 1 Cycle 3 - Not at all: number analyzed (Participants) | 88 | 184
  Day 1 Cycle 3 - Not at all | 43.2 | 46.7
  Day 1 Cycle 3 - A little: number analyzed (Participants) | 88 | 184
  Day 1 Cycle 3 - A little | 45.5 | 41.8
  Day 1 Cycle 3 - Quite a bit: number analyzed (Participants) | 88 | 184
  Day 1 Cycle 3 - Quite a bit | 10.2 | 8.7
  Day 1 Cycle 3 - Very much: number analyzed (Participants) | 88 | 184
  Day 1 Cycle 3 - Very much | 1.1 | 2.7
  Day 1 Cycle 4 - Not at all: number analyzed (Participants) | 82 | 169
  Day 1 Cycle 4 - Not at all | 48.8 | 46.7
  Day 1 Cycle 4 - A little: number analyzed (Participants) | 82 | 169
  Day 1 Cycle 4 - A little | 36.6 | 36.1
  Day 1 Cycle 4 - Quite a bit: number analyzed (Participants) | 82 | 169
  Day 1 Cycle 4 - Quite a bit | 14.6 | 15.4
  Day 1 Cycle 4 - Very much: number analyzed (Participants) | 82 | 169
  Day 1 Cycle 4 - Very much | 0 | 1.8
  Day 1 Cycle 5 - Not at all: number analyzed (Participants) | 64 | 136
  Day 1 Cycle 5 - Not at all | 56.3 | 55.9
  Day 1 Cycle 5 - A little: number analyzed (Participants) | 64 | 136
  Day 1 Cycle 5 - A little | 35.9 | 36.0
  Day 1 Cycle 5 - Quite a bit: number analyzed (Participants) | 64 | 136
  Day 1 Cycle 5 - Quite a bit | 7.8 | 5.9
  Day 1 Cycle 5 - Very much: number analyzed (Participants) | 64 | 136
  Day 1 Cycle 5 - Very much | 0 | 2.2
  Day 1 Cycle 6 - Not at all: number analyzed (Participants) | 59 | 122
  Day 1 Cycle 6 - Not at all | 54.2 | 49.2
  Day 1 Cycle 6 - A little: number analyzed (Participants) | 59 | 122
  Day 1 Cycle 6 - A little | 37.3 | 40.2
  Day 1 Cycle 6 - Quite a bit: number analyzed (Participants) | 59 | 122
  Day 1 Cycle 6 - Quite a bit | 8.5 | 8.2
  Day 1 Cycle 6 - Very much: number analyzed (Participants) | 59 | 122
  Day 1 Cycle 6 - Very much | 0 | 2.5
  Day 1 Cycle 8 - Not at all: number analyzed (Participants) | 48 | 96
  Day 1 Cycle 8 - Not at all | 62.5 | 58.3
  Day 1 Cycle 8 - A little: number analyzed (Participants) | 48 | 96
  Day 1 Cycle 8 - A little | 33.3 | 37.5
  Day 1 Cycle 8 - Quite a bit: number analyzed (Participants) | 48 | 96
  Day 1 Cycle 8 - Quite a bit | 4.2 | 4.2
  Day 1 Cycle 10 - Not at all: number analyzed (Participants) | 42 | 81
  Day 1 Cycle 10 - Not at all | 66.7 | 54.3
  Day 1 Cycle 10 - A little: number analyzed (Participants) | 42 | 81
  Day 1 Cycle 10 - A little | 28.6 | 44.4
  Day 1 Cycle 10 - Quite a bit: number analyzed (Participants) | 42 | 81
  Day 1 Cycle 10 - Quite a bit | 4.8 | 1.2
  Day 1 Cycle 12 - Not at all: number analyzed (Participants) | 36 | 70
  Day 1 Cycle 12 - Not at all | 63.9 | 50.0
  Day 1 Cycle 12 - A little: number analyzed (Participants) | 36 | 70
  Day 1 Cycle 12 - A little | 30.6 | 45.7
  Day 1 Cycle 12 - Quite a bit: number analyzed (Participants) | 36 | 70
  Day 1 Cycle 12 - Quite a bit | 5.6 | 4.3
  Day 1 Cycle 14 - Not at all: number analyzed (Participants) | 31 | 60
  Day 1 Cycle 14 - Not at all | 61.3 | 53.3
  Day 1 Cycle 14 - A little: number analyzed (Participants) | 31 | 60
  Day 1 Cycle 14 - A little | 25.8 | 45.0
  Day 1 Cycle 14 - Quite a bit: number analyzed (Participants) | 31 | 60
  Day 1 Cycle 14 - Quite a bit | 12.9 | 1.7
  Day 1 Cycle 16 - Not at all: number analyzed (Participants) | 28 | 53
  Day 1 Cycle 16 - Not at all | 60.7 | 56.6
  Day 1 Cycle 16 - A little: number analyzed (Participants) | 28 | 53
  Day 1 Cycle 16 - A little | 28.6 | 35.8
  Day 1 Cycle 16 - Quite a bit: number analyzed (Participants) | 28 | 53
  Day 1 Cycle 16 - Quite a bit | 10.7 | 7.5
  Day 1 Cycle 18 - Not at all: number analyzed (Participants) | 23 | 50
  Day 1 Cycle 18 - Not at all | 69.6 | 58.0
  Day 1 Cycle 18 - A little: number analyzed (Participants) | 23 | 50
  Day 1 Cycle 18 - A little | 30.4 | 36.0
  Day 1 Cycle 18 - Quite a bit: number analyzed (Participants) | 23 | 50
  Day 1 Cycle 18 - Quite a bit | 0 | 6.0
  Day 1 Cycle 20 - Not at all: number analyzed (Participants) | 21 | 44
  Day 1 Cycle 20 - Not at all | 71.4 | 59.1
  Day 1 Cycle 20 - A little: number analyzed (Participants) | 21 | 44
  Day 1 Cycle 20 - A little | 28.6 | 31.8
  Day 1 Cycle 20 - Quite a bit: number analyzed (Participants) | 21 | 44
  Day 1 Cycle 20 - Quite a bit | 0 | 9.1
  Day 1 Cycle 22 - Not at all: number analyzed (Participants) | 18 | 36
  Day 1 Cycle 22 - Not at all | 55.6 | 52.8
  Day 1 Cycle 22 - A little: number analyzed (Participants) | 18 | 36
  Day 1 Cycle 22 - A little | 38.9 | 36.1
  Day 1 Cycle 22 - Quite a bit: number analyzed (Participants) | 18 | 36
  Day 1 Cycle 22 - Quite a bit | 5.6 | 11.1
  Day 1 Cycle 24 - Not at all: number analyzed (Participants) | 16 | 34
  Day 1 Cycle 24 - Not at all | 75.0 | 55.9
  Day 1 Cycle 24 - A little: number analyzed (Participants) | 16 | 34
  Day 1 Cycle 24 - A little | 25.0 | 38.2
  Day 1 Cycle 24 - Quite a bit: number analyzed (Participants) | 16 | 34
  Day 1 Cycle 24 - Quite a bit | 0 | 5.9
  Day 1 Cycle 26 - Not at all: number analyzed (Participants) | 15 | 31
  Day 1 Cycle 26 - Not at all | 73.3 | 51.6
  Day 1 Cycle 26 - A little: number analyzed (Participants) | 15 | 31
  Day 1 Cycle 26 - A little | 26.7 | 41.9
  Day 1 Cycle 26 - Quite a bit: number analyzed (Participants) | 15 | 31
  Day 1 Cycle 26 - Quite a bit | 0 | 6.5
  Day 1 Cycle 28 - Not at all: number analyzed (Participants) | 14 | 23
  Day 1 Cycle 28 - Not at all | 64.3 | 56.5
  Day 1 Cycle 28 - A little: number analyzed (Participants) | 14 | 23
  Day 1 Cycle 28 - A little | 35.7 | 39.1
  Day 1 Cycle 28 - Quite a bit: number analyzed (Participants) | 14 | 23
  Day 1 Cycle 28 - Quite a bit | 0 | 4.3
  Day 1 Cycle 30 - Not at all: number analyzed (Participants) | 13 | 20
  Day 1 Cycle 30 - Not at all | 69.2 | 70.0
  Day 1 Cycle 30 - A little: number analyzed (Participants) | 13 | 20
  Day 1 Cycle 30 - A little | 30.8 | 25.0
  Day 1 Cycle 30 - Quite a bit: number analyzed (Participants) | 13 | 20
  Day 1 Cycle 30 - Quite a bit | 0 | 5.0
  Day 1 Cycle 32 - Not at all: number analyzed (Participants) | 12 | 22
  Day 1 Cycle 32 - Not at all | 50.0 | 59.1
  Day 1 Cycle 32 - A little: number analyzed (Participants) | 12 | 22
  Day 1 Cycle 32 - A little | 41.7 | 36.4
  Day 1 Cycle 32 - Quite a bit: number analyzed (Participants) | 12 | 22
  Day 1 Cycle 32 - Quite a bit | 8.3 | 4.5
  Day 1 Cycle 34 - Not at all: number analyzed (Participants) | 11 | 20
  Day 1 Cycle 34 - Not at all | 72.7 | 65.0
  Day 1 Cycle 34 - A little: number analyzed (Participants) | 11 | 20
  Day 1 Cycle 34 - A little | 27.3 | 35.0
  Day 1 Cycle 36 - Not at all: number analyzed (Participants) | 11 | 20
  Day 1 Cycle 36 - Not at all | 63.6 | 65.0
  Day 1 Cycle 36 - A little: number analyzed (Participants) | 11 | 20
  Day 1 Cycle 36 - A little | 36.4 | 35.0
  Day 1 Cycle 38 - Not at all: number analyzed (Participants) | 11 | 18
  Day 1 Cycle 38 - Not at all | 72.7 | 61.1
  Day 1 Cycle 38 - A little: number analyzed (Participants) | 11 | 18
  Day 1 Cycle 38 - A little | 27.3 | 33.3
  Day 1 Cycle 38 - Quite a bit: number analyzed (Participants) | 11 | 18
  Day 1 Cycle 38 - Quite a bit | 0 | 5.6
  Day 1 Cycle 40 - Not at all: number analyzed (Participants) | 11 | 18
  Day 1 Cycle 40 - Not at all | 72.7 | 55.6
  Day 1 Cycle 40 - A little: number analyzed (Participants) | 11 | 18
  Day 1 Cycle 40 - A little | 27.3 | 38.9
  Day 1 Cycle 40 - Quite a bit: number analyzed (Participants) | 11 | 18
  Day 1 Cycle 40 - Quite a bit | 0 | 5.6
  Day 1 Cycle 42 - Not at all: number analyzed (Participants) | 8 | 18
  Day 1 Cycle 42 - Not at all | 75.0 | 66.7
  Day 1 Cycle 42 - A little: number analyzed (Participants) | 8 | 18
  Day 1 Cycle 42 - A little | 25.0 | 33.3
  Day 1 Cycle 44 - Not at all: number analyzed (Participants) | 8 | 16
  Day 1 Cycle 44 - Not at all | 75.0 | 68.8
  Day 1 Cycle 44 - A little: number analyzed (Participants) | 8 | 16
  Day 1 Cycle 44 - A little | 25.0 | 31.3
  Day 1 Cycle 46 - Not at all: number analyzed (Participants) | 8 | 17
  Day 1 Cycle 46 - Not at all | 87.5 | 76.5
  Day 1 Cycle 46 - A little: number analyzed (Participants) | 8 | 17
  Day 1 Cycle 46 - A little | 0 | 23.5
  Day 1 Cycle 46 - Quite a bit: number analyzed (Participants) | 8 | 17
  Day 1 Cycle 46 - Quite a bit | 12.5 | 0
  Day 1 Cycle 48 - Not at all: number analyzed (Participants) | 7 | 14
  Day 1 Cycle 48 - Not at all | 100 | 71.4
  Day 1 Cycle 48 - A little: number analyzed (Participants) | 7 | 14
  Day 1 Cycle 48 - A little | 0 | 28.6
  Day 1 Cycle 50 - Not at all: number analyzed (Participants) | 7 | 11
  Day 1 Cycle 50 - Not at all | 100 | 63.6
  Day 1 Cycle 50 - A little: number analyzed (Participants) | 7 | 11
  Day 1 Cycle 50 - A little | 0 | 36.4
  Day 1 Cycle 52 - Not at all: number analyzed (Participants) | 6 | 10
  Day 1 Cycle 52 - Not at all | 100 | 60.0
  Day 1 Cycle 52 - A little: number analyzed (Participants) | 6 | 10
  Day 1 Cycle 52 - A little | 0 | 40.0
  Day 1 Cycle 54 - Not at all: number analyzed (Participants) | 3 | 8
  Day 1 Cycle 54 - Not at all | 100 | 50.0
  Day 1 Cycle 54 - A little: number analyzed (Participants) | 3 | 8
  Day 1 Cycle 54 - A little | 0 | 50.0
  Day 1 Cycle 56 - Not at all: number analyzed (Participants) | 2 | 3
  Day 1 Cycle 56 - Not at all | 100 | 0
  Day 1 Cycle 56 - A little: number analyzed (Participants) | 2 | 3
  Day 1 Cycle 56 - A little | 0 | 100
  Day 1 Cycle 58 - Not at all: number analyzed (Participants) | 1 | 2
  Day 1 Cycle 58 - Not at all | 100 | 50.0
  Day 1 Cycle 58 - A little: number analyzed (Participants) | 1 | 2
  Day 1 Cycle 58 - A little | 0 | 50.0
  Day 1 Cycle 60 - Not at all: number analyzed (Participants) | 1 | 1
  Day 1 Cycle 60 - Not at all | 100 | 0
  Day 1 Cycle 60 - A little: number analyzed (Participants) | 1 | 1
  Day 1 Cycle 60 - A little | 0 | 100
  Day 1 Cycle 62 - Not at all: number analyzed (Participants) | 1 | 1
  Day 1 Cycle 62 - Not at all | 100 | 0
  Day 1 Cycle 62 - A little: number analyzed (Participants) | 1 | 1
  Day 1 Cycle 62 - A little | 0 | 100
  Day 1 Cycle 64 - A little: number analyzed (Participants) | 0 | 1
  Day 1 Cycle 64 - A little |  | 100

22. Secondary Outcome: Part 2: Percentage of Participants With Ant-Drug Antibodies (ADAs) to Atezolizumab After SC or IV Administration
Description: The percentage of ADA-positive participants after atezolizumab administration was reported. Participants who received atezolizumab were considered to be treatment-emergent ADA-positive if they were ADA-negative or had missing data at baseline but developed an ADA response following atezolizumab exposure (treatment-induced ADA response), or if they were ADA-positive at baseline and the titer of one or more post-baseline samples was at least 0.60 titer units (t.u.) greater than the titer of the baseline sample (treatment-enhanced ADA response). Percentages have been rounded to one decimal place.
Time Frame: From Cycle 1 Day 1 (Cycle length = 21 days) up to treatment discontinuation visit (Up to approximately 20 months)
Population: Safety-evaluable population included all participants who received at least one dose of atezolizumab (IV or SC), with participants grouped according to treatment received. Overall number analyzed is the number of participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Atezolizumab IV 1200 mg | Part 2: Atezolizumab SC 1875 mg
Number analyzed (Participants) | 112 | 228
percentage of participants | 14.3 | 20.6

23. Secondary Outcome: Part 2: Percentage of Participants With ADAs to rHuPH20 After SC Administration
Description: The percentage of ADA-positive participants after atezolizumab SC formulated with rHuPH20 administration was reported. Participants who received atezolizumab SC formulated with rHuPH20 were considered to be treatment-emergent ADA-positive if they were ADA-negative or had missing data at baseline but developed an ADA response following rHuPH20 exposure (treatment-induced ADA response), or if they were ADA-positive at baseline and the titer of one or more post-baseline samples was at least 0.60 t.u. greater than the titer of the baseline sample (treatment-enhanced ADA response). Percentages have been rounded to one decimal place.
Time Frame: From Cycle 1 Day 1 (Cycle length = 21 days) up to treatment discontinuation visit (Up to approximately 20 months)
Population: Safety-evaluable population included all participants who received at least one dose of atezolizumab SC formulated with rHuPH20. Overall number analyzed is the number of participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: Atezolizumab SC 1875 mg
Number analyzed (Participants) | 228
percentage of participants | 5.7

24. Secondary Outcome: Part 2: Percentage of Health Care Professionals (HCPs) by Their Response to Question 2 of HCP SC Versus IV Perspective Questionnaire
Description: The HCP SC versus IV Perspective Questionnaire consisted of five items evaluating the number of atezolizumab SC and IV administrations done, convenience, potential time savings, and overall satisfaction with atezolizumab SC and atezolizumab IV, as well as reasons for HCP-reported satisfaction or dissatisfaction. HCPs who administered at least three doses of atezolizumab as an IV infusion and as a SC injection across all participants in Part 2 of this study responded to this questionnaire, of which question 2 is being reported here: Question 2: Which formulation of atezolizumab (SC or IV) do you think is more convenient for you? Responses to this question are reported in the data table. HCPs were allowed to complete the questionnaire until the last participant completed their assessments (duration between the 'first participant in [FPI]' date to 'last participant last visit [LPLV]' for Part 2).
Time Frame: After HCP has completed administering at least 3 doses of atezolizumab SC and IV across all participants in Part 2 (Up to approximately 48 months)
Population: Overall number analyzed included HCPs who completed Question 2 of the questionnaire.
Measure: Number; unit: percentage of HCPs
Groups:
- Part 2: Atezolizumab IV/Atezolizumab SC: Participants received atezolizumab, 1200 mg, as an IV infusion, Q3W, or atezolizumab, 1875 mg, co-formulated with rHuPH20, as SC injection, on Day 1 of each cycle (1 cycle=21 days) until PD, loss of clinical benefit, or unacceptable toxicity. HCPs who administered the IV or SC formulations completed the HCP SC versus IV Perspective Questionnaire.
Arm/Group | Part 2: Atezolizumab IV/Atezolizumab SC
Number analyzed (Participants) | 50
percentage of HCPs
  Atezolizumab SC is much more convenient | 24.0
  Atezolizumab SC is a little more convenient | 16.0
  Both formulations are equally convenient | 26.0
  Atezolizumab IV is a little more convenient | 12.0
  Atezolizumab IV is much more convenient | 22.0

25. Secondary Outcome: Part 2: Percentage of HCPs by Their Response to Question 3 of the HCP SC Versus IV Perspective Questionnaire
Description: The HCP SC versus IV Perspective Questionnaire consisted of five items evaluating the number of atezolizumab SC and IV administrations done, convenience, potential time savings, and overall satisfaction with atezolizumab SC and atezolizumab IV, as well as reasons for HCP-reported satisfaction or dissatisfaction. HCPs who administered at least three doses of atezolizumab as an IV infusion and as a SC injection across all participants in Part 2 of this study responded to this questionnaire, of which question 3 is being reported here: Question 3: If used in routine practice, do you think administering atezolizumab SC could save staff time compared to atezolizumab IV? The responses to this question could be Yes; No; Unsure. HCPs were allowed to complete the questionnaire until the last participant completed their assessments (duration between the 'FPI in' date to 'LPLV' for Part 2).
Time Frame: as for outcome 24
Population: Overall number analyzed included HCPs who completed Question 3 of the questionnaire.
Measure: Number; unit: percentage of HCPs
Arm/Group | Part 2: Atezolizumab IV/Atezolizumab SC
Number analyzed (Participants) | 50
percentage of HCPs
  Yes | 74.0
  Unsure | 14.0
  No | 12.0

26. Secondary Outcome: Part 2: Percentage of HCPs by Their Response to Question 4 of the HCP SC Versus IV Perspective Questionnaire
Description: The HCP SC versus IV Perspective Questionnaire consisted of five items evaluating the number of atezolizumab SC and IV administrations done, convenience, potential time savings, and overall satisfaction with atezolizumab SC and atezolizumab IV, as well as reasons for HCP-reported satisfaction or dissatisfaction. HCPs who administered at least three doses of atezolizumab as an IV infusion and as a SC injection across all participants in Part 2 of this study responded to this questionnaire, of which question 4 is being reported here: Question 4: Overall, were you more satisfied with atezolizumab SC or atezolizumab IV? The responses included: More satisfied with atezolizumab SC; Equally satisfied with both formulations; More satisfied with atezolizumab IV. HCPs were allowed to complete the questionnaire until the last participant completed their assessments (duration between the 'FPI in' date to 'LPLV' for Part 2).
Time Frame: as for outcome 24
Population: Overall number analyzed included HCPs who completed Question 4 of the questionnaire.
Measure: Number; unit: percentage of HCPs
Arm/Group | Part 2: Atezolizumab IV/Atezolizumab SC
Number analyzed (Participants) | 50
percentage of HCPs
  More satisfied with atezolizumab SC | 32.0
  Equally satisfied with both formulations | 38.0
  More satisfied with atezolizumab IV | 30.0

27. Secondary Outcome: Part 2: Percentage of HCPs by Their Response to Question 2 of the HCP SC Perspective Questionnaire
Description: The HCP SC Perspective Questionnaire consisted of five items evaluating the convenience, ease of administration and overall satisfaction with atezolizumab SC, as well as reasons for HCP-reported satisfaction or dissatisfaction. HCPs who administered at least three doses of atezolizumab as a SC injection across all participants in Part 2 of this study responded to this questionnaire, of which question 2 is being reported here: Question 2: Do you think atezolizumab SC is convenient? The responses to this question could be: Yes; No; and Unsure. HCPs were allowed to complete the questionnaire until the last participant completed their assessments (duration between the 'FPI in' date to 'LPLV' for Part 2). Percentages have been rounded to one decimal place.
Time Frame: After HCP has completed administering at least 3 doses of atezolizumab SC across all participants in Part 2 (Up to approximately 48 months)
Population: Overall number analyzed included HCPs who completed Question 2 of the questionnaire.
Measure: Number; unit: percentage of HCPs
Groups:
- Part 2: Atezolizumab SC 1875 mg: Participants received atezolizumab, 1875 mg, co-formulated with rHuPH20, as SC injection, on Day 1 of each cycle (1 cycle=21 days) until PD, loss of clinical benefit, or unacceptable toxicity. HCPs who administered the SC formulation completed the HCP SC Perspective Questionnaire.
Arm/Group | Part 2: Atezolizumab SC 1875 mg
Number analyzed (Participants) | 84
percentage of HCPs
  Yes | 78.6
  Unsure | 14.3
  No | 7.1

28. Secondary Outcome: Part 2: Percentage of HCPs by Their Response to Question 3 of the HCP SC Perspective Questionnaire
Description: The HCP SC Perspective Questionnaire consisted of five items evaluating the convenience, ease of administration and overall satisfaction with atezolizumab SC, as well as reasons for HCP-reported satisfaction or dissatisfaction. HCPs who administered at least three doses of atezolizumab as a SC injection across all participants in Part 2 of this study responded to this questionnaire, of which question 3 is being reported here: Question 3: Overall, how easy did you find atezolizumab SC administration? The responses to this question could be: Very easy; Fairly easy; Not at all easy. HCPs were allowed to complete the questionnaire until the last participant completed their assessments (duration between the 'FPI in' date to 'LPLV' for Part 2). Percentages have been rounded to one decimal place.
Time Frame: as for outcome 27
Population: Overall number analyzed included HCPs who completed Question 3 of the questionnaire.
Measure: Number; unit: percentage of HCPs
Arm/Group | Part 2: Atezolizumab SC 1875 mg
Number analyzed (Participants) | 84
percentage of HCPs
  Very easy | 54.8
  Fairly easy | 34.5
  Not at all easy | 10.7

29. Secondary Outcome: Part 2: Percentage of HCPs by Their Response to Question 4 of the HCP SC Perspective Questionnaire
Description: The HCP SC Perspective Questionnaire consisted of five items evaluating the convenience, ease of administration and overall satisfaction with atezolizumab SC, as well as reasons for HCP-reported satisfaction or dissatisfaction. HCPs who administered at least three doses of atezolizumab as a SC injection across all participants in Part 2 of this study responded to this questionnaire, of which question 4 is being reported here: Question 4: Overall, how satisfied were you with atezolizumab SC? The responses to this question could be: Very satisfied; Satisfied; Dissatisfied; Very dissatisfied. HCPs were allowed to complete the questionnaire until the last participant completed their assessments (duration between the 'FPI in' date to 'LPLV' for Part 2). Percentages have been rounded to one decimal place.
Time Frame: as for outcome 27
Population: Overall number analyzed included HCPs who completed Question 4 of the questionnaire.
Measure: Number; unit: percentage of HCPs
Arm/Group | Part 2: Atezolizumab SC 1875 mg
Number analyzed (Participants) | 84
percentage of HCPs
  Very satisfied | 34.5
  Satisfied | 50.0
  Dissatisfied | 13.1
  Very dissatisfied | 2.4

ADVERSE EVENTS:
Time Frame: From initiation of the study treatment up to approximately 69 months in Part 1 and up to approximately 44.7 months in Part 2
Description: Safety-evaluable population=all participants who received at least one dose of atezolizumab (IV or SC), with participants grouped according to treatment received.
  HCPs who administered study treatment to participants were not enrolled in the study. To evaluate the HCPs' reported experience with administration of atezolizumab SC & IV, they were asked to complete 2 questionnaires: HCP SC Versus IV Perspective & HCP SC Perspective. No adverse event data were collected for the HCPs in this study.
Arm/Group | Part 1 Cohort 1: Atezolizumab SC Co-mix 1800 mg | Part 1 Cohort 2: Atezolizumab SC Co-mix 1200 mg | Part 1 Cohort 3: Atezolizumab SC Co-mix 1800 mg | Part 2: Atezolizumab IV 1200 mg | Part 2: Atezolizumab SC 1875 mg
All-Cause Mortality (participants affected / at risk) | 4/13 | 6/15 | 19/39 | 97/124 | 206/247
Serious Adverse Events (participants affected / at risk) | 2/13 | 4/15 | 8/39 | 35/124 | 50/247
Other Adverse Events (participants affected / at risk) | 13/13 | 12/15 | 31/39 | 91/124 | 204/247
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Cohort 1: Atezolizumab SC Co-mix 1800 mg (N=13) | Part 1 Cohort 2: Atezolizumab SC Co-mix 1200 mg (N=15) | Part 1 Cohort 3: Atezolizumab SC Co-mix 1800 mg (N=39) | Part 2: Atezolizumab IV 1200 mg (N=124) | Part 2: Atezolizumab SC 1875 mg (N=247)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Autoimmune myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Enteritis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 6 (7) | 8 (8)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Cohort 1: Atezolizumab SC Co-mix 1800 mg (N=13) | Part 1 Cohort 2: Atezolizumab SC Co-mix 1200 mg (N=15) | Part 1 Cohort 3: Atezolizumab SC Co-mix 1800 mg (N=39) | Part 2: Atezolizumab IV 1200 mg (N=124) | Part 2: Atezolizumab SC 1875 mg (N=247)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 5 (8) | 13 (16) | 21 (30) | 47 (54)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 3 (4)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 8 (9)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 7 (7) | 9 (18)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 7 (7)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 1 (1) | 7 (9) | 21 (25)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 12 (12)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 9 (9) | 17 (17)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 1 (1) | 4 (6) | 3 (4) | 21 (27)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (7)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 9 (12) | 4 (4) | 15 (16)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 7 (7)
Asthenia (General disorders) | 5 (5) | 3 (3) | 7 (12) | 9 (11) | 19 (19)
Chest pain (General disorders) | 0 (0) | 1 (2) | 2 (3) | 9 (9) | 11 (14)
Chills (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (2) | 3 (3) | 11 (14) | 16 (20) | 31 (33)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injection site inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 3 (3) | 1 (1) | 2 (4) | 0 (0) | 5 (15)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 5 (5)
Pain (General disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 4 (4)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 1 (1) | 6 (8) | 12 (16)
Xerosis (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (4) | 1 (1) | 3 (3)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 10 (11) | 19 (19)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (4)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 13 (15)
Respiratory tract infection (Infections and infestations) | 1 (5) | 0 (0) | 1 (2) | 2 (3) | 4 (4)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0) | 3 (3) | 3 (3) | 7 (7)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (2) | 1 (1) | 8 (11) | 11 (15)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 5 (9)
Lack of injection site rotation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 5 (5) | 10 (12) | 24 (25)
Amylase increased (Investigations) | 0 (0) | 2 (2) | 5 (6) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 4 (5) | 13 (14) | 23 (28)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 4 (4) | 7 (7) | 20 (21)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 2 (4) | 2 (9) | 1 (2)
Blood cholesterol increased (Investigations) | 1 (3) | 3 (3) | 5 (8) | 1 (2) | 3 (3)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 3 (4) | 7 (8) | 6 (8)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 6 (6) | 12 (16)
Blood magnesium decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Blood sodium decreased (Investigations) | 0 (0) | 2 (2) | 4 (5) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 7 (15)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 7 (7)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (5) | 2 (3) | 5 (6) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 3 (4) | 1 (4) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 2 (2) | 2 (2) | 6 (7) | 15 (18)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 8 (8) | 15 (16) | 31 (32)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (9) | 2 (3)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (10) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3) | 13 (22) | 12 (18)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (4) | 11 (15) | 9 (14)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 5 (6) | 14 (15)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 6 (9) | 8 (9)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 4 (4) | 8 (9) | 8 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 7 (7) | 13 (17) | 17 (18)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 7 (10) | 7 (8) | 18 (21)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3) | 5 (5) | 9 (9) | 21 (21)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 3 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 4 (6) | 11 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (7) | 13 (17)
Hair follicle tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 5 (5) | 5 (6)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 7 (7) | 17 (21)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Sensory loss (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 5 (5)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 8 (8) | 8 (8)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 0 (0) | 1 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (3) | 7 (10) | 9 (9) | 33 (37)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 5 (5) | 20 (21) | 26 (27)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3) | 3 (3) | 7 (9)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 5 (6)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 5 (5)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (7) | 12 (13) | 14 (14)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 10 (14) | 13 (15)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 4 (5) | 3 (10) | 3 (5)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT03735121/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT03735121/SAP_001.pdf